CLINICAL TRIAL: NCT07136571
Title: Phase I Study of Safety and Feasibility of Transarterial Embolization of Incurable Hypervascular Pediatric Soft Tissue Sarcomas
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Junaid Yasin Raja, Assistant Professor, Division of Interventional Radiology, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R25-117; Radiology Research Pilot Award (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2025-08-08; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Soft Tissue Sarcomas
Keywords: TRANSARTERIAL EMBOLIZATION; pediatric; soft tissue sarcoma; incurable
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Pediatric soft tissue sarcoma group (Experimental): Transarterial Embolization
  Interventions: Device: bland particles

INTERVENTIONS:
Device: bland particles — embolization with bland particles of appropriate size
  Other Names: Embozene Color-Advanced Microspheres

SUMMARY:
This is a single center, single arm phase I clinical trial exploring the feasibility and safety of performing transarterial embolization of incurable hypervascular pediatric soft tissue sarcomas with at least an index tumor with 50% arterial enhancement and a 3mm feeding vessel on pre study evaluation. The target study sample size is 10 tumors in a requisite number of participants. These patients will be enrolled to undergo evaluation of all angiographically visible tumors >3cm with subsequent bland (not adsorbed to radioactive or chemotherapy) particle embolization of at least 25% perfusion to the target tumor.

DETAILED DESCRIPTION:
The study will include a screening period in which patient eligibility is determined. Once enrolled parents and patients over 5 years of age will complete a quality-of-life survey PedsQL with a dedicated cancer module and visual analog scale questions for pain and procedural satisfaction. Approximately 2 weeks later the patient will undergo angiography and embolization where feasible. The patient will return for a post-procedural clinic visit at 2-weeks post intervention to assess for adverse effects and complete a follow up PedsQL and VAS surveys. If a major safety event is identified an independent reviewer will review all interim procedures to assess whether excess adverse events have occurred, and the study should be terminated. If this is exceeded the study will be aborted. The patient and parents will also complete PedsQL and VAS surveys in weeks 12- and 24-weeks post intervention. Follow up Computerized Tomography (CT) or Magnetic Resonance Imaging (MRI) concordant with baseline imaging modality will also be performed at weeks 12 and 24 to assess tumoral response.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patient aged 2-18 years, weighing at least 20 kg
* Diagnosed with biopsy proven primary or metastatic soft tissue sarcoma designated as a non-curative surgical candidate and/or failure of standard of care chemotherapy/immunotherapy with local progression on 3-month post induction imaging
* Staging CT or MRI demonstrating at least 50% arterial vascularity by volume within at least one tumor measuring at least 3 cm in longest dimension with an identifiable arterial feeder within one month of screening visit

Exclusion Criteria:

* Negative pregnancy test within 48 hours of angiography or lactation for females of childbearing age
* Known anaphylactic allergic reactions to iodinated contrast
* Planned surgery or radiation to the target site within the study period at time of enrollment

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Rate of technical success will be defined as proportion of enrolled patients that were able to undergo angioembolization of at least 25% of the target tumor by volume as determined by post-procedure cone beam CT imaging. | procedure/surgery
  Safety will be evaluated by the number of patients with non-pain related major adverse events according to the Common Terminology Criteria for Adverse Events (CTCAE) criteria.
  The study population to be explored no longer fits within a defined standard of care protocol. These patients unfortunately have a poor overall life expectancy and have not had a positive response to existing medication and radiation protocols. Transarterial embolization may offer a palliative treatment modality with potential benefit to patients in this cohort provided that it may be able to be performed successfully and safely. The minimal clinical acceptance performance standard for transarterial tumor embolization in the target population is 50% and will serve as the comparator for the primary outcome measure of percent of enrolled patients achieving technical procedural success.

SECONDARY OUTCOMES:
Local disease control will be assessed on 3- and 6-month staging MRI or CT scans using modified Response Evaluation Criteria in Solid Tumors (mRECIST) criteria. | Baseline to 6 months
  Local disease control for these patients who otherwise do not have a standard of care protocol may offer palliation or potential survival benefit as has been seen in other, mostly adult, cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Junaid Raja, MD, MSPH, FACP, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No